CLINICAL TRIAL: NCT03002077
Title: An Open-label, Long-term Safety Study of Rapastinel as Adjunctive Therapy in Patients With Major Depressive Disorder
Brief Title: Long-term Safety Study of Rapastinel as Adjunctive Therapy in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAP-MD-06
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Results first posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — GLYX-13 peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rapastinel (Experimental): Rapastinel 450 milligrams (mg) intravenous (IV) open label weekly or every two weeks, based on investigator's discretion for 52 Weeks.
  Interventions: Drug: Rapastinel

INTERVENTIONS:
Drug: Rapastinel — Rapastinel pre-filled syringes for IV injections.

SUMMARY:
This study will evaluate the long-term safety and tolerability of rapastinel as an adjunctive to antidepressant therapy (ADT) in patients with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for MDD
* Current major depressive episode of at least 8 weeks and not exceeding 18 months in duration at Screening
* Have no more than partial response (< 50% improvement) to ongoing treatment with a protocol-allowed antidepressant
* If female of childbearing potential, have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test.

Exclusion Criteria:

* DSM-5-based diagnosis of any disorder other than MDD that was the primary focus of treatment within 6 months before Screening
* Lifetime history of meeting DSM-5 criteria for:
* Schizophrenia spectrum or other psychotic disorder
* Bipolar or related disorder
* Major neurocognitive disorder
* Neurodevelopmental disorder of greater than mild severity or of a severity that impacts the participant's ability to consent, follow study directions, or otherwise safely participate in the study
* Dissociative disorder
* Posttraumatic stress disorder
* MDD with psychotic features
* Significant suicide risk, as judged by the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Hoogerheyde, Study Director — Allergan
Locations (128):
- United States (128):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Harmonex, Inc., Dothan, Alabama
  - NoesisPharma, Phoenix, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - California Pharmaceutical Research Institute, Inc, Anaheim, California
  - Southern California Research LLC., Beverly Hills, California
  - ATP Clinical Research Inc., Costa Mesa, California
  - ProScience Research Group, Culver City, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Sun Valley Research Center, Imperial, California
  - Irvine Center for Clinical Research, Inc, Irvine, California
  - Synergy Clinical Research Center of Escondido, Lemon Grove, California
  - Synergy San Diego, Lemon Grove, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pacific Research Partners; LLC., Oakland, California
  - Excell Research, Oceanside, California
  - NRC Research Institute, Orange, California
  - Asclepes Research Centers, Panorama City, California
  - Anderson Clinical Research, Redlands, California
  - CITrials, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - PCSD Feighner Research, San Diego, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - Thomas M. Shiovitz, M.D., Inc., DBA California Neuroscience Research Medical Group, Inc.,, Sherman Oaks, California
  - Viking Clinical Research, Temecula, California
  - Pacific Clinical Research Medical, Upland, California
  - MCB Clinical Research Center, Colorado Springs, Colorado
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Meridien Research, Bradenton, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - MD Clinical, Hallandale, Florida
  - Reliable Clinical Research, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Meridien Research, Lakeland, Florida
  - Innovative Clinical Research, Inc, Lauderhill, Florida
  - Innova Clinical Trials Inc., Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - Research Centers of America, Oakland Park, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Combined Research Orlando Phase I-IV, Orlando, Florida
  - Millenia Psychiatry & Research, Inc, Orlando, Florida
  - Olympian Clinical Research, Tampa, Florida
  - University of South Florida, Psychiatry and Behavioral Neurosciences, Tampa, Florida
  - Institute for Advanced Medical Research, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Iris Research, Smyrna, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - AMR - Baber Research, Inc., Naperville, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Louisiana Clinical Research, Shreveport, Louisiana
  - J Gary Booker, MD APMC, Shreveport, Louisiana
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Pharmasite Research, Inc, Baltimore, Maryland
  - CBH Health, Gaithersburg, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices & Research, Inc., Methuen, Massachusetts
  - Coastal Research Associates, South Weymouth, Massachusetts
  - Adams Clinical Trials, Watertown, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Millennium Psychiatric Associates, St Louis, Missouri
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Altea Research, Las Vegas, Nevada
  - Healthy Perspectives - Innovative Mental Health Services. PLLC, Nashua, New Hampshire
  - Hassman Research Institute, LLC, Berlin, New Jersey
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Pharmaceutical Research Associates Inc, Marlton, New Jersey
  - Global Medical Institute, LLC, Princeton, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Neuroscience, Inc, Albuquerque, New Mexico
  - SPRI Clinical Trials, Inc, Brooklyn, New York
  - Bioscience Research, Mount Kisco, New York
  - Manhattan Behavioral Medicine, New York, New York
  - Eastside Comprehensive Medical Center, LLC, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Fieve Clinical Research, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Carolina Clinical Trials, Inc., Charleston, North Carolina
  - New Hope Clinical Research Inc., Charlotte, North Carolina
  - Richard H. Weisler, MD, PA, Raleigh, North Carolina
  - Neuro-Behavioral Clinical Research, Inc, Canton, Ohio
  - Patient Priority Clinical Site, LLC, Cincinnati, Ohio
  - The Ohio State University Department of Psychiatry, Columbus, Ohio
  - Midwest Clinical Research Center LLC, Dayton, Ohio
  - Charak Clinical Research Center, Garfield Heights, Ohio
  - Lindner Center of Hope, Mason, Ohio
  - Professional Psychiatric Services, Mason, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - Red River Medical Research Center, LLC, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Inc, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, Oklahoma City, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - Coastal Carolina Research Center, Inc., Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - Donald J. Garcia, Jr., MD, PA, Austin, Texas
  - Community Clinical Research, Inc., Austin, Texas
  - BioBehavioral Research of Austin, Austin, Texas
  - Houston Clinical Trials, LLC, Bellaire, Texas
  - Relaro Medical Trials, Dallas, Texas
  - El Campo Clinical Trials, El Campo, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Earle Research, Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Family Psychiatry of The Wood, The Woodlands, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Psychiatric and Behavioral Solutions, Salt Lake City, Utah
  - Pharmaceutical Research Associates, Inc, Salt Lake City, Utah
  - Psychiatric Alliance of the Blue Ridge, Inc., Charlottesville, Virginia
  - NorthWest Clinical Research Center, Bellevue, Washington
  - Pacific Institute of Medical Sciences, Bothell, Washington

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned to be terminated when 100 patients had completed the 52-week Open Label Treatment Period (OLTP).
Pre-assignment Details: Patients who either completed the RAP-MD-04 Double-blind Treatment Period (DBTP) or who did not meet criteria to be randomized into the DBTP of RAP-MD-04 and were therefore discontinued from that study were eligible for Study RAP-MD-06.
Period: Overall Study
Arm/Group | Rapastinel
Started | 617
Completed | 179
Not Completed | 438
Not completed — Non-compliance with Study Drug | 4
Not completed — Non-compliance w/Background ADT | 1
Not completed — Study Terminated by Sponsor | 257
Not completed — Site Terminated by Sponsor | 5
Not completed — Miscellaneous Reasons | 10
Not completed — Adverse Event | 23
Not completed — Lack of Efficacy | 20
Not completed — Withdrawal by Subject | 72
Not completed — Lost to Follow-up | 21
Not completed — Pregnancy | 4
Not completed — Protocol Violation | 21

BASELINE CHARACTERISTICS:
Population: The Safety Population consisted of all screened patients who received at least 1 dose of rapastinel during the OLTP of the study.
Arm/Group | Rapastinel
Number analyzed (Participants) | 617
Age, Continuous [Median (Standard Deviation); unit: Years] | 46.5 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 455
  Male | 162
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 83
  Not Hispanic or Latino | 534
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 485
  Black or African American | 107
  Asian | 12
  American Indian or Alaska Native | 2
  Native Hawaiian or Other Pacific Islander | 4
  Multiple | 7

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: 52 Weeks
Population: as for baseline characteristics
Measure: Number; unit: Count of Participants
Arm/Group | Rapastinel
Number analyzed (Participants) | 617
Count of Participants | 457

2. Secondary Outcome: Change From Baseline in Brief Psychiatric Rating Scale Positive Symptoms Subscale (BPRS+)
Description: The BPRS+ is a subset of the BPRS that assesses 4 components of the BPRS+ related to the degree of psychosis: Conceptual Disorganization, Suspiciousness, Hallucinatory Behavior, and Unusual Thought Content assessed by the investigator using a 7-point scale ranging from 1=Not Present to 7=Extremely Severe for a total possible score of 0 (best) to 28 (worst). A negative change from Baseline indicates improvement.
Time Frame: Baseline to 52 Weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rapastinel
Number analyzed (Participants) | 617
Scores on a scale | -0.0 (0.33)

3. Secondary Outcome: Change From Baseline in the Clinician Administered Dissociative States Scale (CADSS)
Description: The Clinician Administered Dissociative States Scale (CADSS) is a clinician-administered measure of perceptual, behavioral, and attentional alterations occurring during active dissociative experiences composed of 23 subjective self-reported and 5 objective observer-reported ratings, each scored from 0 (not at all) to 4 (extremely). Only the 23 subjective items will be collected and analyzed. The sum of each of the 23 subjective items was used for a total score of 0-92. A negative change from Baseline indicates improvement.
Time Frame: Baseline to 52 Weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Rapastinel
Number analyzed (Participants) | 617
Scores on a Scale | -0.2 (1.24)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected up to 52 weeks during the OLTP.
Description: The Safety Population consisted of all screened patients who received at least 1 dose of rapastinel during the OLTP of the study.
Arm/Group | Rapastinel
All-Cause Mortality (participants affected / at risk) | 0/617
Serious Adverse Events (participants affected / at risk) | 28/617
Other Adverse Events (participants affected / at risk) | 285/617
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Rapastinel (N=617)
Suicidal ideation (Psychiatric disorders) | 4
Major depression (Psychiatric disorders) | 2
Abortion induced (Surgical and medical procedures) | 1/455
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/455
Abscess jaw (Infections and infestations) | 1
Accelerated hypertension (Vascular disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Alcohol use disorder (Psychiatric disorders) | 1
Appendiceal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Appendicitis perforated (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Depression (Psychiatric disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/455
Epstein-Barr virus infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Gastroenteritis (Infections and infestations) | 1
Gun shot wound (Infections and infestations) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1
Presyncope (Nervous system disorders) | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1
Renal failure (Renal and urinary disorders) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Transient ischaemic attack (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rapastinel (N=617)
Upper respiratory tract infection (Infections and infestations) | 89
Nasopharyngitis (Infections and infestations) | 78
Headache (Nervous system disorders) | 71
Dysgeusia (Nervous system disorders) | 43
Nausea (Gastrointestinal disorders) | 43
Back pain (Musculoskeletal and connective tissue disorders) | 37
Insomnia (Psychiatric disorders) | 36
Weight increased (Investigations) | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-06-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT03002077/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT03002077/SAP_001.pdf